CLINICAL TRIAL: NCT05730881
Title: Comparison of Four Intensive Care Scores in Prediction of Survival After Veno-Arterial ECMO: A Single Center Retrospective Study
Brief Title: Comparison of Four Intensive Care Scores in Prediction of VA-ECMO Survival.
Acronym: ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-22-701
Record Dates: First submitted 2022-12-05; First posted 2023-02-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-11

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation Complication
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ECMO — VA-ECMO is a life support measures, we need to estimate the survival by different techniques to allocate therapeutic interventions properly

SUMMARY:
VA-ECMO is increasingly utilized in the setting of cardiogenic shock or cardiac arrest to restore hemodynamic stability and end organ function. VA-ECMO serves as a short-term ventricular assist device that can be rapidly placed at the bedside in the emergency room, intensive care unit, cardiac catheterization suite, or operating room. A bridge to decision approach allows for the assessment of neurologic status, renal and hepatic function, and subsequent recovery of cardiac function. Despite its life-saving potential, VA-ECMO is fraught with complications including vascular complications from cannulation. In addition, neurologic injury, renal failure, liver failure, and sepsis are all well described sequelae of the post-cardiogenic shock or cardiac arrest VA-ECMO patient. For these reasons, identifying early prognostic indicators and developing a score with regard to the outcome of this special patient population is of high interest. The proposed study aims to analyze 4 ICU scores/Survival prediction models [APACHE-II (acute physiology and chronic health evaluation II), SAVE (Survival after VA ECMO) , SOFA (sequential organ failure assessment )and CASUS (Cardiac Surgery Score)] and evaluate their performance in predicting survival after VA ECMO insertion. This will be a clinical retrospective study which will be conducted in the Cardiothoracic Intensive Care unit (CTICU) in the Department of Cardiothoracic Surgery, Heart Hospital, Doha. Patients admitted to the CTICU after institution of VA ECMO in the period between 1st January 2015 to 31st October 2022 will be screened retrospectively. Patients who stay for at least 12 hours in the CTICU would be eligible for inclusion in the study. All charts of patients who were admitted to CTICU after institution of VA ECMO during the afore mentioned period will be included in the review. All the risk scores would be calculated separately for all the enrolled patients and then subjected to statistical analysis to determine predictive accuracy for survival.

ELIGIBILITY:
* Inclusion criteria

  * Age more than18 years old.
  * Patients undergoing institution of VA ECMO
* Exclusion criteria

  * Patients staying < 12 hours in the ICU

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be undertaken in the Cardiothoracic intensive care unit (CTICU) in the Heart hospital, Hamad Medical Corporation for patients who require VA-ECMO support
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Survival predictive accuracy of four scores | 6 months
  Survival predictive accuracy of four scores

CONTACTS AND LOCATIONS:
Overall Officials: Suraj Sudarsanan, Md, Principal Investigator — Hamad medical coproation
Locations (1):
- Hamad medical corporation, Doha, DA, Qatar